CLINICAL TRIAL: NCT04489615
Title: DELTA-CAPNO: Identification of Risk Factors for Alteration of the Cellular-arterial Gradient of CO2 in Pre-hospital Patients
Brief Title: Identification of Risk Factors for Alteration of the Cellular-arterial Gradient of CO2
Acronym: DELTA-CAPNO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: UH Angers
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Mechanical Ventilation; Prehospital Capnography Monitoring
Keywords: capnography prehospital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Monocentric, prospective, observational and descriptive study on the evaluation of risk factors for alteration of the alveoarterial gradient of CO2 in pre-hospital patients, intubated and then ventilated in an invasive manner; and their impact on intra-arterial fatehospital.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age,
* Endotracheal intubation in pre-hospital and mechanical ventilation,
* Monitoring of Etco2 in pre-hospital settings

Exclusion Criteria:

* Identification of a chest wound blowing during pre-hospital care,
* No technical possibility for performing or analysing arterial sampling,
* Death during pre-hospital care,
* A person who has objected to the processing of his data for research at minimal risk and constraints (category 2) or for research on data, as well as persons subject to legal protection measures.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included are the major patients, intubated and ventilated in pre-hospital, transferred by the medical team to the University Hospital of Angers.
  The ventilation settings are left to the caregiver's discretion, as is the purpose of Etco2.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
identification of risks factors for alteration of the cellular arterial gradient of CO2 in Pre hospital patients | from january 2020 to april 2021
  The main objective is therefore to determine the main risk factors to observe an alteration of the alveoarterial gradient in CO2, at the hospital care (fixed at 10 mmHg).

SECONDARY OUTCOMES:
Intrahospital mortality | from january 2020 to april 2021
  prognostic evidence of altered alveocapillary gradient on intrahospital mortality
Time of hospital admission | from january 2020 to april 2021
  the prognosis of the finding of an altered alveocapillary gradient on the time of hospital admission
length of mecanical ventilation | from january 2020 to april 2021
  the prognosis of the finding of an altered alveocapillary gradient on the duration of ventilation
Occurence of pneumonia | from january 2020 to april 2021
  the prognosis of the finding of an altered alveocapillary gradient on the occurrence of pneumonia
Acute respiratory distress syndrom (ARDS) | from january 2020 to april 2021
  the prognosis of the finding of an altered alveocapillary gradient on the occurrence of ARDS
Length of stay | from january 2020 to april 2021
  the prognosis of the finding of an altered alveocapillary gradient on the length of stay
Intrahospital mortality (subpopulation of traumatized patients which had suffered from intracranial hypertension | from january 2020 to april 2021
  prognostic evidence of altered alveocapillary gradient, onset of an episode of intracranial hypertension, and intrahospital survival of severely traumatized patients (GCS < 9).

CONTACTS AND LOCATIONS:
Overall Officials: Quentin qc Carraro, md, Principal Investigator — UH Angers
Locations (1):
- Quentin Carraro, Angers, France

IPD SHARING:
Plan to Share IPD: No